CLINICAL TRIAL: NCT05806645
Title: UPTAKE: Using Personalized Risk and Digital Tools to Guide Transitions Following Acute Kidney Events- A Pragmatic Randomized Controlled Trial in Connect Care
Brief Title: UPTAKE: Using Personalized Risk and Digital Tools to Guide Transitions Following Acute Kidney Events
Acronym: UPTAKE-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other); Canadian Institutes of Health Research (CIHR) (Other Government); University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UPTAKE Pro00128939
Record Dates: First submitted 2023-03-22; First posted 2023-04-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: This is a waiver of consent trial, participants will be randomized to an enhanced discharge care pathway vs usual care in the electronic health record.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The proposed experimental intervention will incorporate our risk prediction model which will be used in combination with a patients medical profile to guide the hospital to home transition of care for low, medium and high-risk groups of patients. Patients will receive transition of care plans that are tailored to their medical profile and embedded within standardized discharge pathways within the electronic health record
  Interventions: Other: Risk-guided transition of care intervention delivered through an integrated digital health strategy
- Usual Care (No Intervention): The usual care group will not receive the risk-guided transition of intervention and will receive standard hospital discharge care in accordance with local health system standards (Alberta Health Services), with recommendations for kidney function, proteinuria and laboratory testing at 90 days after discharge.

INTERVENTIONS:
Other: Risk-guided transition of care intervention delivered through an integrated digital health strategy — Patients will receive transition of care plans that are tailored to their medical profile and risk and embedded within standardized discharge pathways within the EHR- Education and self-management guidance about AKI for patients, Medication guidance based on evidence-based indications for reducing risk of cardiac and kidney outcomes, Recommendations for subsequent laboratory testing of kidney function, proteinuria and electrolytes according to clinical characteristics and risks, Recommendations for timing and nature of PCP follow-up, Information about the patient's AKI and subsequent management provided to PCPs through discharge summary, Recommendations for outpatient Pharmacy follow-up for medication reconciliation and review according to patient risk and medication management gaps, Recommendations for Nephrology referral for high risk patients
  Arms: Intervention

SUMMARY:
Nearly one in ten people who are hospitalized in Canada develop a complication with sudden loss of kidney function, called acute kidney injury (AKI). AKI may lead to other severe health problems after discharge home, such as kidney failure requiring dialysis treatment, heart failure, heart attacks, stroke, and even premature death. Discharge from hospital to home can be a difficult transition where there are often gaps in identification, communication, care coordination, education, and planning of care for AKI. The study team will co-design and evaluate a tailored post-discharge care plan that is based on the risk of later kidney problems and uses currently available, yet untapped digital innovation to improve the health and experience of people with AKI.

This study will be built into Alberta's new Epic Systems based provincial electronic health record (EHR). The plan is to use digital tools in the EHR to identify all people in Alberta hospitals that have had an AKI event and are at increased risk of long-term complications. Half will randomly be assigned to receive a tailored care plan based on their risk at hospital discharge while the other half will receive care as it is currently provided by their healthcare team. The electronic health system will automatically calculate a patient's risk and report this risk in their chart along with recommendations for care. The study team includes patients, healthcare providers, and health system decision makers needed to co-develop the proposed strategy and introduce the changes needed to deliver this intervention. The investigators will study whether this strategy can reduce health problems that may happen after AKI including death, chronic kidney disease (CKD), kidney failure, heart attacks, and stroke. The investigators will also determine if the approach improves patient experience during the transition from hospital to home. This study has the potential to revolutionize how we care for people that leave hospital after having AKI.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is common in hospitalized patients and associated with poor long-term outcomes including kidney failure, cardiovascular (CV) events, and death, with highest risk in older adults. The transition of hospitalized patients with AKI to home is challenging, with many care gaps. Identifying those at highest risk of adverse post-discharge outcomes and delivering interventions to reduce the risk of progressive kidney and CV disease via appropriate, acceptable, and efficient intervention strategies are needed. Our team has developed and externally validated a risk prediction model for hospitalized adults with AKI, which can estimate the risk of advanced chronic kidney disease (eGFR<30mL/min/1.73m2 or kidney failure). The investigators used this risk model to guide follow-up in a pilot trial for AKI survivors within Alberta (ClinicalTrials.gov: NCT02915575). The investigators have found that a risk-guided strategy to follow-up is a feasible approach to close gaps in care; however, larger studies are required to evaluate broader implementation, and impact on patient-centered outcomes, costs, and sustainability in a real-world setting. Alberta Health Services (AHS) has implemented a new province-wide clinical information system which provides a unique opportunity to use digital health technology to design and evaluate a risk-guided hospital-to-home transition of care intervention that builds upon previous work.

OBJECTIVES AND METHODS:

1. To co-develop a risk-guided intervention with patients, clinicians, and health system decision-makers to improve personalized transitions of care between hospital and home for survivors of AKI. The investigators will use a participatory research approach that engages patients and care providers to co-design an evidence-guided, experience-based intervention for AKI transitions in care. Qualitative methods will be used to identify and prioritize transition interventions aligned with patient risk of adverse post-discharge outcomes.
2. To a) identify key service delivery supports required to integrate the AKI hospital to home transition of care intervention and b) establish usability and acceptability of the intervention within the electronic health record. With the support of the AHS and existing hospital to home transition initiatives, the investigators will work with key health system partners to integrate developed AKI transition of care intervention within the EHR. The investigators will use a mixed methods approach to identify barriers and enablers to implementation and establish usability and acceptability of the intervention.
3. To evaluate the effectiveness of this intervention in a pragmatic clinical trial that will measure implementation success and impact on patient experience, outcomes, and costs. Using the EHR, hospitalized adults with AKI at increased risk of adverse long-term outcomes will be randomized to the risk-guided transition intervention or usual care. The risk-guided arm will receive the interventions identified in Objective 1 tailored based on their clinical profile and risk of CKD from the prediction model. The primary outcome of the trial is the two-year risk of a composite of death, kidney failure, or major CV event. 6,046 patients are required to detect a 15% relative risk reduction of the primary outcome, with 90% power. Effects on patient experience, processes of care, implementation, and costs will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

(all of)

* Age ≥ 18 years old
* Hospitalized at site using AHS EHR
* Acute Kidney Injury (Stage 1-3) identified in hospital per KDIGO guideline criteria

Exclusion Criteria:

(any of)

* Pre-hospitalization advanced CKD: eGFR<30 mL/min/1.73m2
* Pre-hospitalization dialysis
* Very low risk (<1% risk) of advanced CKD
* Non-Alberta resident
* Palliative goals of care
* Enrolled in the UPTAKE VC Trial
* Admitted under a nephrologist at time of discharge
* Dialysis on at least 2 days in the last week prior to discharge
* Receiving apheresis
* Kidney transplant recipient
* Diagnosis of Glomerulonephritis
* Cirrhosis AND complication of cirrhosis in medical history or active problem list (ascites, varices, hepatic encephalopathy, hepatorenal syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6046 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Primary effectiveness outcome | 2 years after discharge
  The primary outcome of the study is major adverse kidney or CV events within 2 years after discharge, defined as the composite of death, kidney failure (receipt of maintenance dialysis, kidney transplant or eGFR < 15 mL/min/1.73m2 for 4 weeks or more), or hospitalization with a most responsible diagnosis for heart failure, myocardial infarction, or stroke (based on validated ICD-10 coding algorithms)

SECONDARY OUTCOMES:
Secondary Clinical Outcomes-Death | 2 years of discharge
  Death from any cause within 2 years of discharge
Safety Outcomes- Hyperkalemia | within 1 year of discharge
  Serum potassium ≥ 6.0 mEq/L on outpatient lab testing within one year of discharge
Safety Outcomes-Hospitalization for Kidney Disease Ambulatory Care Specific Condition | within 1 year of discharge
  Hospitalization for a Kidney Disease Ambulatory Care Specific Condition (Congestive Heart Failure, Volume Overload, Hyperkalemia, or Hypertensive Emergency) within one year after discharge (based on ICD-10 coding algorithms)
Safety Outcomes-All Cause Hospitalization or ED Visit | 30 and 90 days of discharge
  All-cause hospitalization or ED visits within 30 and 90 days of discharge
Secondary Clinical Outcomes-Kidney Failure | within 2 years of discharge
  Receipt of maintenance dialysis, kidney transplant, or eGFR < 15 mL/min/1.73m2 for 4 weeks or more) within 2 year of discharge
Secondary Clinical Outcomes-Hospitalization for CV Events | Within 2 years of hospital discharge
  Hospitalization with a most responsible diagnosis for heart failure, myocardial infarction, or stroke (based on validated ICD-10 coding algorithms) within 2 years of hospital discharge
Patient Experience | 3 months post discharge
  Patient experience will be assessed using a survey with six questions related to AKI transition in care administered by AHS via phone 3 months post discharge to a random estimated 10% of patients in both control and intervention arms of the study. The sampling frame will be designed to recruit an equal number of patients from each CKD risk strata.
Implementation Outcomes | 2 or 4 weeks of discharge
  Implementation outcomes will include the proportion of eligible patients included in the study who receive each element of the enhanced care intervention that is recommended by the practice advisory, according to their risk strata. These will include documentation of AKI in the problem list, AKI discharge communication sent to the patient's primary care provider at discharge, after visit summary printed for the patient prior to discharge, referral to community pharmacist when recommended, referral to nephrologist when recommended, and laboratory test (eGFR, urine ACR, electrolytes) ordered for within 2 or 4 weeks of discharge according to recommendations.
Process of Care Outcomes | within 2 or 4 weeks or 90 days of discharge
  Process of care outcomes will include the proportion of patients who receive the recommended kidney function monitoring (eGFR, urine ACR, electrolytes) within 2 or 4 weeks after discharge, the proportion of patients with a recommendation for and who receive a guideline-indicated medication for kidney and cardiovascular risk reduction (RAAS blockers, SGLT-2 inhibitors, finerenone, and statin prescription) within 90 days of discharge, the proportion of patients reviewed by a community pharmacist within 4 weeks when recommended, and the proportion of patients seen by a nephrologist within 4 weeks when recommended.

CONTACTS AND LOCATIONS:
Overall Officials: Neesh Pannu, Principal Investigator — University of Alberta; Matthew James, Principal Investigator — University of Calgary; Tyrone Harrison, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No